CLINICAL TRIAL: NCT02923401
Title: High-Intensity Interval Training for Women at Heightened Risk for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0442; NCI-2016-01938 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Disorders of Breast
Keywords: Exercise; Biomarkers; Breast cancer high risk; Treadmill; Stationary bicycle; Questionnaires; Surveys; Motivational sessions; Phone calls; Printed materials
MeSH Terms: conditions — Breast Diseases; Motor Activity | interventions — Exercise; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-Intensity Interval Training (HIIT) Group (Experimental): Participants come to the Energy Balance Center to exercise 3 times a week for 12 weeks.
  Participants receive written materials and instructions on how to perform their exercises.
  Participants walk uphill on a treadmill for a total of 33 minutes 3 times a week for 12 weeks.
  Participants complete questionnaires about their quality of life, exercise experience, and level of fatigue at baseline and at 12 weeks.
  One (1) time each month, participant attends a motivational session.
  Interventions: Other: Exercise; Behavioral: Questionnaires; Behavioral: Motivational Session; Other: Printed Materials
- Moderate-Intensity Continuous Training (MICT) Group (Experimental): Participants come to the Energy Balance Center to exercise 3 times a week for 12 weeks.
  Participants receive written materials and instructions on how to perform their exercises.
  Participants walk uphill on a treadmill or use a stationary bicycle continuously for 41 minutes 3 times a week for 12 weeks.
  Participants complete questionnaires about their quality of life, exercise experience, and level of fatigue at baseline and at 12 weeks.
  One (1) time each month, participant attends a motivational session.
  Interventions: Other: Exercise; Behavioral: Questionnaires; Behavioral: Motivational Session; Other: Printed Materials
- Control Group (Active Comparator): Participants receive written materials and counseling by an exercise physiologist.
  Participants called by a member of the study staff 1 time each week for 12 weeks and asked about any exercise they have done and their weight loss goals.
  Participants complete questionnaires about their quality of life, exercise experience, and level of fatigue at baseline and at 12 weeks.
  One (1) time each month, participant attends a motivational session.
  Interventions: Behavioral: Questionnaires; Behavioral: Motivational Session; Behavioral: Phone Call

INTERVENTIONS:
Other: Exercise — High-Intensity Interval Training (HIIT) Group: Participants walk uphill on a treadmill for a total of 33 minutes 3 times a week for 12 weeks.There is a 5-minute warm up, followed by four 4-minute intervals. Between each interval, participant walks for 3 minutes. There is a 3 minute cool down.
  Moderate-Intensity Continuous Training (MICT) Group: Participants walk uphill on a treadmill or use a stationary bicycle continuously for 41 minutes 3 times a week for 12 weeks.
  Arms: High-Intensity Interval Training (HIIT) Group; Moderate-Intensity Continuous Training (MICT) Group
Behavioral: Questionnaires — Participants complete questionnaires about their quality of life, exercise experience, and level of fatigue at baseline and at 12 weeks. These should take a total of about 15 minutes to complete.
  Other Names: Surveys
Behavioral: Motivational Session — One (1) time each month, participant attends a motivational session for 12 weeks.
Behavioral: Phone Call — Participants called by a member of the study staff 1 time each week for 12 weeks and asked about any exercise they have done and their weight loss goals. Each phone call should take about 15 minutes.
  Arms: Control Group
Other: Printed Materials — High-Intensity Interval Training (HIIT) Group and Moderate-Intensity Continuous Training (MICT) Group: Participants receive written materials and instructions on how to perform their exercises.
  Control Group: Participants receive written materials and counseling by an exercise physiologist.
  Arms: High-Intensity Interval Training (HIIT) Group; Moderate-Intensity Continuous Training (MICT) Group

SUMMARY:
The goal of this research study is to learn if there is a level of exercise training that is more effective in lowering biomarker levels that are linked to breast cancer risk. Biomarkers are found in the blood/tissue and may be related to your reaction to exercise.

This is an investigational study. Up to 72 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Groups:

If you agree to take part in this research study, you will be randomly assigned (as in a roll of dice) to 1 of 3 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance of being assigned to each group:

* If you are in Group 1, you will take part in high-intensity interval (HIIT) exercise.
* If you are in Group 2, you will take part in moderate-intensity exercise.
* If you are in Group 3, you will not take part in any assigned exercise, but you will receive written materials and counseling by an exercise physiologist.

If you are in Group 1 or Group 2, you will also receive written materials and instructions on how to perform your exercises.

Physical Activity:

If you are in Group 1 or 2, you will come to the Energy Balance Center to exercise 3 times a week for 12 weeks.

If you are in Group 1, you will walk uphill on a treadmill for a total of 33 minutes. There will be a 5-minute warm up, followed by four 4-minute intervals. Between each interval, you will walk for 3 minutes. There will be a 3 minute cool down.

If you are in Group 2, you will exercise at the Energy Balance Center 3 times a week. You will walk uphill on a treadmill or use a stationary bicycle continuously for 41 minutes.

If you are in Group 3, 1 time each month while you are on study, you will be called by a member of the study staff and asked about any exercise you have done and your weight loss goals. Each phone call should take about 15 minutes.

The exercise training intensity may be reduced or stopped temporarily if you experience side effects.

Length of Study:

No matter which group you are in, your participation in this study will be over after 12 weeks. You will be taken off study if you have intolerable side effects.

Study Visits:

All participants will visit the MD Anderson Behavioral Research and Treatment Center for each study visit.

At baseline:

* You will have a cardiopulmonary exercise test (CPET) to check your lung function. The CPET checks how well your lungs are working by measuring how much oxygen and carbon dioxide your lungs take in and release when you breathe. To perform this test, you will be asked to walk on a treadmill until you reach a point that you can no longer exercise. You will be breathing into the machine while you walk. This test will take about 30 minutes to complete. The study doctor will be present for each CPET and available to respond to any complication.
* You will have an EKG to check your heart function. The study doctor will be present for each EKG you have.
* Blood (about 1½ tablespoons) will be drawn for biomarker testing. You will be asked to fast (eat nothing and drink only water) for at least 12 hours before each blood draw as part of this study.
* You will have a dual-energy x-ray absorptiometry (DEXA) scan to measure your body mass.
* You will complete a questionnaire that will ask you about your demographics (age, race, and so on), past medical history, and lifestyle habits. This questionnaire should take about 5 minutes to complete.
* You will complete 5 questionnaires about your quality of life, exercise experience, and level of fatigue. These should take a total of about 15 minutes to complete.

At 6 weeks:

* You will have a CPET.
* You will have an EKG.

At 12 weeks:

* You will have a CPET.
* Blood (about 1½ tablespoons) will be drawn for biomarker testing.
* You will have an EKG.
* You will have a DEXA scan.
* You will complete the same questionnaires that you completed at baseline.
* If you are in Group 1 or 2, you will be interviewed by a member of the study staff. You will be asked 5 questions about your experience with your assigned exercise program. It should take about 5 minutes to complete.

One (1) time each month, you will attend a motivational session. During this session, you will discuss strategies for overcoming barriers that may be keeping you from attending or completing your exercises. You will also talk about continuing physical activity after you complete the program. This session should last about 15-30 minutes.

Additional Information:

* Trained health professionals will be present at all study visits to address any symptoms during exercise. If you feel that you are having difficulty breathing, experiencing dizziness, or are having any heart related symptoms while exercising at home, please stop exercising and call 911 immediately.
* Clinical information such as your name, patient medical record number, age, gender, body mass index (BMI), zip code, and your complete medical history will be collected from your medical record.
* If you are in Group 1 or Group 2, you will receive text messages before each exercise session to remind you to attend. You will be responsible for any text messaging charges. Standard text message rates will apply.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women [defined per provider discretion and notated in the medical record]
2. At high risk of developing breast cancer (history of Ductal Carcinoma In Situ (DCIS), Lobular Carcinoma In Situ (LCIS), Atypical Ductal Hyperplasia (ADH), Gail 5 year risk > 1.66% or lifetime risk > 20%)
3. Enrolled on the Longitudinal High Risk Cohort study or being seen in the Cancer Prevention Center.
4. Oriented to person, place, and time
5. BMI > or equal to 25 kg/m2
6. Speaks and reads English

Exclusion Criteria:

1. Underlying medical problems that contraindicate unsupervised exercise.
2. Women with a prior history of cardiovascular disease, defined as a 1 or more positive responses on the Heart Questionnaire (Appendix D).
3. Uses a walker or wheelchair/scooter
4. Is being treated for diagnosed diabetes or autoimmune disease
5. Lives outside the greater Houston area (Harris and contiguous counties)
6. Is pregnant (self-reported)
7. Is taking risk reduction therapy such as tamoxifen
8. Participants with a blood pressure >=140/90 at the time of baseline testing.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of High-Intensity Interval Exercise to Offset the Tumor Promoting Effects of Obesity in High-Risk Breast Cancer Participants | 12 weeks
  Trials judged feasible if:
  At least 45% of screened patients meet inclusion criteria, 2. At least 50% of patients who meet the inclusion criteria consent, 3. Adherence in HIIT and MICT is larger than 80%, and 4. Retention rate is larger than 80%.

CONTACTS AND LOCATIONS:
Overall Officials: Susan C. Gilchrist, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Coletta AM, Agha NH, Baker FL, Niemiro GM, Mylabathula PL, Brewster AM, Bevers TB, Fuentes-Mattei E, Basen-Engquist K, Gilchrist SC, Simpson RJ. The impact of high-intensity interval exercise training on NK-cell function and circulating myokines for breast cancer prevention among women at high risk for breast cancer. Breast Cancer Res Treat. 2021 Jun;187(2):407-416. doi: 10.1007/s10549-021-06111-z. Epub 2021 Feb 8. PMID 33555464
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org